CLINICAL TRIAL: NCT04812951
Title: Cyclosporine 0.1% Eye Drops as Prophylactic Treatment in Post Surgical Ocular Surface System Failure Within The Age
Brief Title: Cyclosporine 0.1% Eye Drops as Prophylactic Treatment In Cataract Surgery
Acronym: CSA2020
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Antonio Di Zazzo, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSA2020
Record Dates: First submitted 2021-03-15; First posted 2021-03-24 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Ocular Surface Disease; Ocular Inflammation
Keywords: ocular surface disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- young control (No Intervention): 25 patients < 65 years old without any prophylactic anti-inflammatory preoperative treatment
- control (No Intervention): 25 patients > 75 years old without any prophylactic anti-inflammatory preoperative treatment
- Study group (Experimental): 25 patients > 75 years old with prophylactic anti-inflammatory preoperative treatment
  Interventions: Drug: CycloSPORINE Ophthalmic 0.1% Ophthalmic Emulsion
- Vehicle group (Active Comparator): 25 patients > 75 years old with vehicle preoperative treatment
  Interventions: Device: cationorm eye drops

INTERVENTIONS:
Drug: CycloSPORINE Ophthalmic 0.1% Ophthalmic Emulsion — one cyclosporine 0.1% eye drop twice a day for 30 preoperative days
  Other Names: Ikervis eye drops
  Arms: Study group
Device: cationorm eye drops — one cationorm eye drop twice a day for 30 preoperative days
  Arms: Vehicle group

SUMMARY:
Use of Cyclosporine 0.1% Eye Drops as Prophylactic Treatment in cataract Surgery

DETAILED DESCRIPTION:
To asses ocular discomfort symptoms and signs and inflammatory biomarkers after preoperative topical cyclosporine 0.1% eye drops therapy in high risk elder population after a specific insult such as cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Postmenopausal women for whom cataract surgery has been scheduled
* Stage N2-3; C1-2 according (Lens Opacities classification System) LOCS
* Willing to sign informed consent and fully participate to all length of the study
* Patients without any previous medical history of ocular and/or systemic inflammatory, autoimmune or auto inflammatory disease
* Patient with no history of ocular surgery
* Patients without any previous or concomitant ocular diseases

Exclusion Criteria:

* Patients under topical or systemic anti- inflammatory drugs Patients with a concomitant diagnosis of glaucoma, or on therapy with antiglaucoma drugs
* Patients on systemic or local therapy with drugs that alter the secretion of the tear film (beta blockers, antidepressants and psychotropics)
* Patients with a history of allergic, congenital, autoimmune systemic diseases
* Patients who have undergone previous eye surgery
* Ocular or peri-ocular malignancies or premalignant conditions
* Active or suspected ocular or peri-ocular infection.
* Complicated Cataract Surgery
* Patients with a positive pregnancy testAllergy or reaction history to study drug
* Patients who participated in a clinical trial in which an investigational drug was administered within 30 days or 5 half-lives of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Symptoms Assessment Questionnaire iN Dry Eye | 4 months
  SANDE (frequency and severity scores; 0-100)
National Eye Institute grading scale | 4 months
  NEI corneal staining ( n/15 score; 0-15)
Rate of tears' production | 4 months
  Schirmer test (mm/5min)
Tears Break Up Time | 4 months
  T-BUT (Seconds)

SECONDARY OUTCOMES:
Biomarkers' expression in conjunctival epithelial cells | 4 months
  HLA DR (molecular expression)
Biomarkers' expression in conjunctival epithelial cells | 4 months
  ICAM-1 (molecular expression)

CONTACTS AND LOCATIONS:
Locations (1):
- University Campus Bio Medico, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
1. Screening visit (-30 days)
  2. Cataract surgery
  3. visit 1 ( 7 days after surgery)
  4. visit 2 (15 days after surgery)
  5. visit 3 (45 days after surgery),
  6. last follow up (90 days after surgery)

REFERENCES:
- [Background] Gupta PK, Drinkwater OJ, VanDusen KW, Brissette AR, Starr CE. Prevalence of ocular surface dysfunction in patients presenting for cataract surgery evaluation. J Cataract Refract Surg. 2018 Sep;44(9):1090-1096. doi: 10.1016/j.jcrs.2018.06.026. Epub 2018 Aug 2. PMID 30078540
- [Background] Kim JS, Lee H, Choi S, Kim EK, Seo KY, Kim TI. Assessment of the Tear Film Lipid Layer Thickness after Cataract Surgery. Semin Ophthalmol. 2018;33(2):231-236. doi: 10.1080/08820538.2016.1208764. Epub 2016 Sep 14. PMID 27627886
- [Background] Trattler WB, Majmudar PA, Donnenfeld ED, McDonald MB, Stonecipher KG, Goldberg DF. The Prospective Health Assessment of Cataract Patients' Ocular Surface (PHACO) study: the effect of dry eye. Clin Ophthalmol. 2017 Aug 7;11:1423-1430. doi: 10.2147/OPTH.S120159. eCollection 2017. PMID 28848324
- [Background] Iglesias E, Sajnani R, Levitt RC, Sarantopoulos CD, Galor A. Epidemiology of Persistent Dry Eye-Like Symptoms After Cataract Surgery. Cornea. 2018 Jul;37(7):893-898. doi: 10.1097/ICO.0000000000001491. PMID 29504953
- [Background] Kohli P, Arya SK, Raj A, Handa U. Changes in ocular surface status after phacoemulsification in patients with senile cataract. Int Ophthalmol. 2019 Jun;39(6):1345-1353. doi: 10.1007/s10792-018-0953-8. Epub 2018 Jun 20. PMID 29926365
- [Background] Kasetsuwan N, Satitpitakul V, Changul T, Jariyakosol S. Incidence and pattern of dry eye after cataract surgery. PLoS One. 2013 Nov 12;8(11):e78657. doi: 10.1371/journal.pone.0078657. eCollection 2013. PMID 24265705
- [Background] Micera A, Di Zazzo A, Esposito G, Longo R, Foulsham W, Sacco R, Sgrulletta R, Bonini S. Age-Related Changes to Human Tear Composition. Invest Ophthalmol Vis Sci. 2018 Apr 1;59(5):2024-2031. doi: 10.1167/iovs.17-23358. PMID 29677365
- [Background] Di Zazzo A, Micera A, De Piano M, Cortes M, Bonini S. Tears and ocular surface disorders: Usefulness of biomarkers. J Cell Physiol. 2019 Jul;234(7):9982-9993. doi: 10.1002/jcp.27895. Epub 2018 Dec 4. PMID 30515814
- [Background] Olivieri F, Prattichizzo F, Grillari J, Balistreri CR. Cellular Senescence and Inflammaging in Age-Related Diseases. Mediators Inflamm. 2018 Apr 17;2018:9076485. doi: 10.1155/2018/9076485. eCollection 2018. No abstract available. PMID 29849499
- [Background] Baker JR, Vuppusetty C, Colley T, Hassibi S, Fenwick PS, Donnelly LE, Ito K, Barnes PJ. MicroRNA-570 is a novel regulator of cellular senescence and inflammaging. FASEB J. 2019 Feb;33(2):1605-1616. doi: 10.1096/fj.201800965R. Epub 2018 Aug 29. PMID 30156909
- [Background] Ventura MT, Casciaro M, Gangemi S, Buquicchio R. Immunosenescence in aging: between immune cells depletion and cytokines up-regulation. Clin Mol Allergy. 2017 Dec 14;15:21. doi: 10.1186/s12948-017-0077-0. eCollection 2017. PMID 29259496
- [Background] Torricelli AA, Santhiago MR, Wilson SE. Topical cyclosporine a treatment in corneal refractive surgery and patients with dry eye. J Refract Surg. 2014 Aug;30(8):558-64. doi: 10.3928/1081597X-20140711-09. PMID 25325897
- [Background] Di Zazzo A, Micera A, Coassin M, Varacalli G, Foulsham W, De Piano M, Bonini S. InflammAging at Ocular Surface: Clinical and Biomolecular Analyses in Healthy Volunteers. Invest Ophthalmol Vis Sci. 2019 Apr 1;60(5):1769-1775. doi: 10.1167/iovs.18-25822. PMID 31022299